CLINICAL TRIAL: NCT03092674
Title: A Randomized Phase II/III Trial of "Novel Therapeutics" Versus Azacitidine in Newly Diagnosed Patients With Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndrome (MDS), Age 60 or Older LEAP: Less-Intense AML Platform Trial
Brief Title: Azacitidine With or Without Nivolumab or Midostaurin, or Decitabine and Cytarabine Alone in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00436; NCI-2017-00436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1612 (Other: SWOG); S1612 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myelodysplastic Syndrome/Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; GATA2 Deficiency | interventions — Azacitidine; Cytarabine; Decitabine; Injections; midostaurin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (azacitidine) (Active Comparator): Patients receive azacitidine SC or IV daily on days 1-7 or on an interrupted schedule which ensures that all 7 days of therapy are received within a 12 day period. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis
- Arm B (azacitidine, nivolumab) (Experimental): Patients receive azacitidine as in Arm A and nivolumab IV over 30-60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Arm C (azacitidine, midostaurin) (Experimental): Patients receive azacitidine as in Arm A and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Midostaurin
- Arm D (decitabine, cytarabine) (Experimental): INDUCTION: Patients receive decitabine IV over 2 hours on days 1-5 and cytarabine IV continuously on days 6-11. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients deemed stable at the discretion of the treating physician receive decitabine as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Decitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm A (azacitidine); Arm B (azacitidine, nivolumab); Arm C (azacitidine, midostaurin)
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm D (decitabine, cytarabine)
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Arm D (decitabine, cytarabine)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Midostaurin — Given PO
  Other Names: CGP 41251; CGP41251; N-Benzoyl-Staurosporine; N-Benzoylstaurosporine; PKC 412; PKC-412; PKC412; Rydapt
  Arms: Arm C (azacitidine, midostaurin)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm B (azacitidine, nivolumab)

SUMMARY:
This randomized phase II/III trial studies how well azacitidine with or without nivolumab or midostaurin, or decitabine and cytarabine alone work in treating older patients with newly diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome. Drugs used in chemotherapy, such as azacitidine, decitabine, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Midostaurin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving azacitidine with or without nivolumab or midostaurin, or decitabine and cytarabine alone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To select, based on overall survival, any or all of the "Novel Therapeutic" regimens for further testing against azacitidine in patients age 60 and older with newly diagnosed acute myeloid leukemia (AML) or myelodysplastic syndrome with excessive blasts-2 (MDS-EB-2). (Phase II) II. To compare overall survival of the "Novel Therapeutic" regimens selected in the phase II portion of the trial to azacitidine in these patient populations. (Phase III)

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities of the regimens in these patient populations.

II. To estimate response rates, event-free survival, and relapse-free survival for these regimens in these patient populations.

TERTIARY OBJECTIVES:

I. To investigate associations between cytogenetic and molecular abnormalities (including FLT3) and outcomes for each of the regimens in these patient populations.

II. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM A: Patients receive azacitidine subcutaneously (SC) or intravenously (IV) daily on days 1-7 or on an interrupted schedule which ensures that all 7 days of therapy are received within a 12 day period. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive azacitidine as in Arm A and nivolumab IV over 30-60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive azacitidine as in Arm A and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM D:

INDUCTION: Patients receive decitabine IV over 2 hours on days 1-5 and cytarabine IV continuously on days 6-11. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients deemed stable at the discretion of the treating physician receive decitabine as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for the 1st year, every 6 months for the 2nd and 3rd years, then annually until 5 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION STEP 1-SPECIMEN SUBMISSION
* Patients must be suspected to have previously untreated acute myelogenous leukemia (AML) or myelodysplastic syndrome with excess blasts-2 (MDS-EB-2)
* Patients must not be known to have AML in the central nervous system (CNS)
* Patients must have specimens submitted for FLT3 testing for randomization stratification; collection of pretreatment specimens must be completed within 1 day of registration to Step 1; specimens must be submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System; FLT3 results will be used for stratification purposes at the time of randomization; E-mail notification of randomization assignment must be received prior to Step 2 registration
* Patients must be offered participation in specimen banking; with patient consent, pretreatment specimens must be collected and submitted via the SWOG Specimen Tracking System
* Patients who have received prior therapy with midostaurin, any anti-PD-1 or anti-PD-L1 therapy, any deoxyribonucleic acid (DNA)-methyltransferase inhibitor (including hypomethylating agents such as azacitidine, decitabine, or other investigational agent that acts by inhibiting DNA or ribonucleic acid [RNA] methylation) for any condition, or prior intensive cytotoxic therapy for myelodysplastic syndrome (MDS), are not eligible
* Patients must be able to swallow oral medications without crushing or chewing
* Prior malignancy is allowed providing it does not require concurrent therapy

  * Exception: active hormonal therapy is allowed
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception also includes (but is not limited to) heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or vasectomy; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

  * Women must agree to avoid breast-feeding and women of child-bearing potential (WOCBP) must agree to use highly effective contraception while receiving study drug and for a period of 31 weeks after the last dose of study drug; sexually-active men must agree to use a condom while receiving study drug and for 31 weeks after the last dose of study drug; vasectomized men must also agree to use a condom to avoid delivering drug in the seminal fluid
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* REGISTRATION STEP 2-RANDOMIZATION: Patients must be registered to Step 2 no more than 42 days after registration to Step 1 and no more than 42 days after collection of specimens for FLT3 testing
* REGISTRATION STEP 2-RANDOMIZATION: Patients must have morphologically confirmed, previously untreated acute myeloid leukemia (AML) or MDS with excess blasts-2 (MDS-EB-2)

  * Patients with acute promyelocytic leukemia (APL), biphenotypic leukemia, blastic transformation of chronic myelogenous leukemia (CML or BCR/ABL), are not eligible
  * Patients must have disease present in the blood or bone marrow; patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible
  * All tests for establishing baseline disease status eligibility must be based on blood and/or bone marrow examination performed within 42 days prior to randomization (registration Step 2)
* REGISTRATION STEP 2-RANDOMIZATION: Patients must not be known to have AML in the CNS
* REGISTRATION STEP 2-RANDOMIZATION: Patients must be deemed, in the judgment of the treating physician, to be ineligible for intensive induction therapy, or must have refused intensive induction therapy; rationale for clinical determination or notation of patient decision must be made
* REGISTRATION STEP 2-RANDOMIZATION: Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 42 days prior to randomization (registration Step 2); reports of the results must be submitted
* REGISTRATION STEP 2-RANDOMIZATION: FLT3 results will be used for stratification purposes at the time of randomization; E-mail notification that FLT3 specimens have been processed must be received prior to randomization (registration Step 2)
* REGISTRATION STEP 2-RANDOMIZATION: Prior treatment with hydroxyurea is permitted; prior all-trans retinoic acid (ATRA) for suspected APL and prior intrathecal therapy are permitted, but must plan to be discontinued prior to initiating protocol therapy; patients with signs/symptoms of hyperleukocytosis or white blood cells (WBC) >= 50,000/mcL can be treated with leukapheresis prior to randomization (registration to Step 2)
* REGISTRATION STEP 2-RANDOMIZATION: Patients may have received non-intensive therapy for antecedent hematologic disorders, including lenalidomide; patients may have received prior chemotherapy for prior cancers; these therapies must be discontinued at least 5 days prior to randomization (registration to Step 2)
* REGISTRATION STEP 2-RANDOMIZATION: Patients who are transfusion-dependent and patients receiving growth factor support are eligible; patients must discontinue growth factor support prior to initiation of protocol therapy
* REGISTRATION STEP 2-RANDOMIZATION: The following tests must be performed within 14 days prior to randomization (registration to Step 2) to establish baseline values:

  * Performance status
  * Complete blood count (CBC)/differential/platelets
  * Creatinine clearance (Cockcroft-Gault)
  * Total bilirubin
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)
  * Lactate dehydrogenase (LDH)
  * Albumin
  * Glucose
  * Fibrinogen
  * Electrocardiogram (ECG)
* REGISTRATION STEP 2-RANDOMIZATION: Patients must have complete history and physical examination within 28 days prior to randomization (registration to Step 2); history must include autoimmune disease status (to determine whether patient is eligible for Arm B)
* REGISTRATION STEP 2-RANDOMIZATION: Patients must not have active infection (systemic bacterial, fungal, or viral infection) that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement despite appropriate antibiotics or other treatment)
* REGISTRATION STEP 2-RANDOMIZATION: Patients must be eligible for at least one of the currently active investigational treatment arms (S1612B or S1612C); if the patient does not meet eligibility criteria for at least one active investigational arm, then the patient is not eligible for S1612
* REGISTRATION STEP 2-RANDOMIZATION: Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* ARM B (AZACITIDINE + NIVOLUMAB)
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients must have AST and ALT =< 2.5 x institutional upper limit of normal (IULN)
* Patients must have total bilirubin =< 1.5 x IULN
* Patients must have baseline troponin test performed for eligibility; however, no associated values must be met in order for the patient to be eligible
* ARM C (AZACITIDINE + MIDOSTAURIN)
* Patients must have total bilirubin =< 2.5 x IULN
* Patients must have creatinine clearance =< 2.5 x IULN
* Patients must have corrected QT (QTc) interval < 500/msec (by Bazett's formula) on baseline ECG
* Patients must not have any history of hypersensitivity to any drugs or metabolites of midostaurin
* All tests for establishing baseline values must be completed within 14 days prior to registration to Step 2 (randomization)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Michaelis, Principal Investigator — SWOG Cancer Research Network
Locations (506):
- United States (506):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - The Watson Clinic, Lakeland, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Medicine Heartland Hematology Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - University of Rochester, Rochester, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 78 participants were initially randomized to the study, 26 per arm. Two were ineligible, one on the Azacitidine+Nivolumab arm and one in the Azacitidine+Midostaurin arm. 76 participants were eligible and included in the primary analysis (26 in the Azacitidine arm, 25 in the Azacitidine+Nivolumab arm, and 25 in the Azacitidine+Midostaurin arm).
Groups:
- Azacitidine: Patients receive azacitidine SC or IV daily on days 1-7 or on an interrupted schedule which ensures that all 7 days of therapy are received within a 12 day period. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Azacitidine + Nivolumab: Patients receive azacitidine as in Arm A and nivolumab IV over 30-60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Azacitidine + Midostaurin: Patients receive azacitidine as in Arm A and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine + Midostaurin
Started | 26 | 25 | 25
Completed | 0 | 0 | 0
Not Completed | 26 | 25 | 25
Not completed — Adverse Event or Side Effects | 1 | 4 | 4
Not completed — Refusal Unrelated to Adverse Event | 5 | 1 | 3
Not completed — Progression/Relapse | 5 | 4 | 8
Not completed — Death | 4 | 8 | 2
Not completed — Other - Not Protocol Specified | 11 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Azacitidine +Midostaurin: Patients receive azacitidine as in Arm A and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin | Total
Number analyzed (Participants) | 26 | 25 | 25 | 76
Age, Continuous [Median (Full Range); unit: years] | 75.5 [61.9 to 86.3] | 76.4 [66.4 to 86.5] | 76.2 [65.7 to 85.8] | 75.6 [61.9 to 86.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 28
  Male | 15 | 17 | 16 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 23 | 23 | 71
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 23 | 21 | 21 | 65
  Race: Black | 2 | 3 | 2 | 7
  Race: Asian | 1 | 0 | 0 | 1
  Race: Unknown | 0 | 1 | 2 | 3
Baseline Blast Percentage [Count of Participants; unit: Participants]
  <20% (MDS-EB-2) | 8 | 5 | 6 | 19
  >=20% (AML) | 18 | 20 | 19 | 57
FLT3-Centrally Reviewed [Count of Participants; unit: Participants]
  Wild Type FLT3-ITD | 25 | 21 | 22 | 68
  Mutated FLT3-ITD | 1 | 4 | 3 | 8
Zubrod Performance Status [Count of Participants; unit: Participants] — Zubrod sacle ranges from 0-4, higher scores reflecting greater disability 0: Fully active, able to carry on all pre-disease performance w/o restriction
  1. Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature, e.g., light housework, office work
  2. Ambulatory & capable of self-care but unable to carry out any work activities; up & about > 50% of waking hours
  3. Capable of limited self-care, confined to bed or chair > 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    0-1 | 21 | 21 | 20 | 62
    2-4 | 5 | 4 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) (Phase II)
Description: Time from date of randomization on study until death from any cause with observations censored on the day of last contact for patients not known to have died.
Time Frame: Day of registration on study until death from any cause, assessed for up to 5 years
Population: The analysis population includes the 76 participants who were eligible and evaluable (26 in the Azacitidine arm, 25 in the Azacitidine+Nivolumab arm, and 25 in the Azacitidine+Midostaurin arm).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
Number analyzed (Participants) | 26 | 25 | 25
months | 6.2 [3.9 to 10] | 5.2 [1.1 to 13.1] | 7.4 [2.9 to 16.4]

2. Primary Outcome: OS (Phase III)
Description: as for outcome 1
Time Frame: Day of registration on study until death from any cause, assessed for up to 5 years
Population: Due to unexpected toxicities on the Azacitidine + Nivolumab arm during the first two cycles of therapy, the trial was closed early, before the phase II portions was completed and before reaching the phase III portion.
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine + Midostaurin
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably, or definitely related to study drugs are reported. CTCAE Version 5.0 was used for all AE reporting.
Time Frame: Duration of treatment and follow up until death or 5 years post randomization (registration to Step 2).
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
Number analyzed (Participants) | 25 | 25 | 23
Participants
  Acidosis | 1 | 0 | 0
  Acute kidney injury | 0 | 1 | 0
  Alanine aminotransferase increased | 0 | 1 | 0
  Anemia | 12 | 10 | 13
  Anorexia | 0 | 0 | 1
  Arthralgia | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Atrial fibrillation | 0 | 0 | 1
  Back pain | 0 | 0 | 1
  Blood and lymphatic system disorders - Other, spec | 1 | 0 | 1
  Cardiac troponin I increased | 1 | 0 | 0
  Catheter related infection | 1 | 0 | 0
  Chest pain - cardiac | 0 | 0 | 1
  Colitis | 0 | 0 | 1
  Constipation | 0 | 1 | 0
  Dry mouth | 0 | 0 | 1
  Dyspnea | 0 | 0 | 1
  Ejection fraction decreased | 0 | 1 | 0
  Electrocardiogram QT corrected interval prolonged | 0 | 0 | 1
  Epistaxis | 1 | 0 | 0
  Fatigue | 1 | 1 | 4
  Febrile neutropenia | 10 | 7 | 8
  Fever | 0 | 1 | 0
  Gastrointestinal disorders - Other, specify | 1 | 0 | 0
  Generalized muscle weakness | 0 | 1 | 1
  Heart failure | 1 | 1 | 2
  Hyperglycemia | 0 | 0 | 1
  Hypertension | 0 | 0 | 1
  Hypoalbuminemia | 1 | 1 | 0
  Hypokalemia | 1 | 1 | 0
  Hyponatremia | 0 | 1 | 1
  Hypophosphatemia | 0 | 1 | 0
  Hypotension | 0 | 2 | 4
  Hypoxia | 1 | 1 | 0
  INR increased | 0 | 0 | 1
  Immune system disorders - Other, specify | 0 | 1 | 0
  Infections and infestations - Other, specify | 0 | 1 | 3
  Joint infection | 0 | 0 | 1
  Lung infection | 2 | 6 | 4
  Lymphocyte count decreased | 3 | 5 | 8
  Mucositis oral | 0 | 0 | 2
  Neutrophil count decreased | 10 | 10 | 15
  Platelet count decreased | 11 | 9 | 10
  Pneumonitis | 0 | 1 | 0
  Pruritus | 1 | 0 | 0
  Pulmonary edema | 0 | 0 | 1
  Rash maculo-papular | 1 | 0 | 0
  Respiratory failure | 0 | 1 | 1
  Sepsis | 2 | 4 | 1
  Skin infection | 0 | 1 | 0
  Small intestinal perforation | 1 | 0 | 0
  Sudden death NOS | 0 | 1 | 0
  Supraventricular tachycardia | 1 | 0 | 0
  Typhlitis | 0 | 0 | 1
  White blood cell decreased | 12 | 10 | 16

4. Other Pre Specified Outcome: Remission Rates
Description: #participants(ps) w comp response(resp)(CR), comp remission w incomp bld ct recovery(CRp/CRi), morphol leukemia-free state(MLFS), erythroid&neutrophil&platelet resp(HI-E,HI-N,HI-P), HI-P, marrow comp resp(CRm), stable disease(SD), no resp(NR) CR:BM blasts<5%; no circ blasts&blasts w Auer rods(AR); no extramedullary disease(ED); ANC≥1x10^9/L; plt ct≥100x10^9/L CRp/CRi:CR criteria excl residual neutropenia<1x10^9/L or ITP<100x10^9/L MLFS:BM blasts<5%; no blasts w AR, ED, hem recovery rqd HI-E:≥1.5g/dL↑Hb pretx;&RBC trans-depen ps, achieve trans independ or relevant↓RBC trans rqd HI-N:ANC↑pretx≥100%,&an absolute↑of>500/mm3 pretx HI-P:Absolute↑≥30000/mm3 pretx for ps w plt ct>20000/mm3 pretx. Ps w plt ct≤20000/mm3 pretx,↑≥100% pretx ct to plt ct>20000/mm3. Plt trans-depend ps, plt trans independ rqd CRm:CR for BM exam≤5%myeloblasts&marrow myeloblasts↓≥50%pretx SD:Not achieve≥PR, w no evidence prog NR:Not achieve CR,CRi,PR,MLFS,SD, excl ps w death in aplasia or due to indet cause
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
Number analyzed (Participants) | 26 | 25 | 25
Participants
  Complete Response | 3 | 4 | 6
  CRp/CRi | 3 | 1 | 0
  MLFS | 1 | 0 | 0
  HI-E and HI-N and HI-P | 1 | 0 | 0
  HI-P only | 0 | 1 | 1
  CRm | 0 | 0 | 1
  Stable disease | 8 | 6 | 7
  No response | 10 | 13 | 10

5. Other Pre Specified Outcome: OS
Description: Will be estimated using the Kaplan-Meier method or Cox regression models. Landmark analyses of different response categories will be evaluated based on dates at which 75% and 90% of patients have achieved a response (with other quantiles analyzed as needed).
Time Frame: Day of registration on study until death from any cause, assessed for up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Relapse-free Survival (RFS)
Description: Time from the date of achievement of a remission (defined as patients achieving complete remission (CR), or CR with incomplete hematological recovery (CRi)) until the date of relapse or death from any cause; patients not known to have relapsed or died at last follow-up are censored on the date of last contact.
Time Frame: Date of achievement of a remission until the date of relapse or death from any cause, assessed for up to 5 years
Population: The analysis population includes the 17 participants who were eligible and evaluable and had complete response or complete remission with incomplete blood count recovery (CRp/CRi) (6 in the Azacitidine arm, 5 in the Azacitidine+Nivolumab arm, and 6 in the Azacitidine+Midostaurin arm).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
Number analyzed (Participants) | 6 | 5 | 6
months | 3.5 [0.6 to 13.3] | 9.4 [1.5 to 17.1] | 13.3 [4 to 26.8]

7. Other Pre Specified Outcome: Event-free Survival (EFS)
Description: Time from from the date of randomization to the first of: date of primary refractory disease; date of progressive disease; date off protocol therapy without CR or CRi; date of relapse from CR or CRi, or death from any cause; patients not known to have any of these events are censored on the date of last contact.
Time Frame: Date of randomization to the first of: date of primary refractory disease; date of progressive disease; date off protocol therapy without CR or CRi; date of relapse from CR or CRi, or death from any cause, assessed for up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
Number analyzed (Participants) | 26 | 25 | 25
months | 3.6 [1.1 to 4.1] | 1.8 [0.6 to 2.7] | 4.5 [1.8 to 9.8]

8. Other Pre Specified Outcome: Cumulative Incidence of Relapse Defined as Achieving CR or CRi
Description: Cumulative incident endpoints and associations will be assessed using Cox regression models (for cause-specific hazards as appropriate).
Time Frame: Date of achievement of a remission until the date of relapse or death, assessed for up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: FLT3-ITD
Description: The prognostic effect of FLT3-ITD (positive versus negative or non-evaluable) with respect to the outcome OS will be evaluated using Cox regression models. The predictive effect of FLT3-ITD (positive versus negative/non-evaluable) with respect to the outcome of OS and the treatments of azacitdine+midostaurin versus azacitidine will be evaluated using a Cox regression model with treatment arm and FLT3-ITD as covariates and including the interaction between the two covariates.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Cytogenetic Abnormalities, Risk Categories, and Mutations in Bone Marrow
Description: Univariate and multivariable regression models will be used to assess potential associations between outcomes (CR, OS, EFS, and RFS) and cytogenetic abnormalities and mutation status (including FLT3-ITD). Regression models including interaction terms with treatment arm will be fit. In addition to analyzing FLT3-ITD as categorical variable used in randomization stratification, we will analyze FLT3-TKD also and evaluate FLT3-ITD allelic ratio as a quantitative variable and as a binary variable using the threshold of 0.50.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Potential Control Arm Drift
Description: Only concurrently randomized patients will be evaluated in comparisons between arms.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post randomization (registration to Step 2).
Description: CTCAE version 5.0 was used for reporting toxicities and SAEs. There were 25 participants in the Azacitidine arm, 25 participants in the Azacitidine + Nivolumab arm, and 23 participants in the Azacitidine + Midostaurin arm that were evaluable for AEs.
Groups:
- Azacitidine: Patients receive azacitidine SC or IV daily on days 1-7 or on an interrupted schedule which ensures that all 7 days of therapy are received within a 12 day period. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. One participant withdrew from protocol therapy before starting treatment and is therefore included in the All-Cause Mortality but not Serious Adverse Events.
- Azacitidine +Midostaurin: Patients receive azacitidine as in Arm A and midostaurin orally (PO) twice daily (BID) on days 8-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. One participant withdrew from protocol therapy before starting treatment and one participant died before starting treatment, therefore these two participants are included in the All-Cause Mortality but not Serious Adverse Events.
Arm/Group | Azacitidine | Azacitidine + Nivolumab | Azacitidine +Midostaurin
All-Cause Mortality (participants affected / at risk) | 24/26 | 25/25 | 23/25
Serious Adverse Events (participants affected / at risk) | 9/25 | 20/25 | 17/23
Other Adverse Events (participants affected / at risk) | 23/25 | 23/25 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=25) | Azacitidine + Nivolumab (N=25) | Azacitidine +Midostaurin (N=23)
Anemia (Blood and lymphatic system disorders) | 2 | 5 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 8 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 4
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 1
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Esophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 2
Death NOS (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 1
Fever (General disorders) | 0 | 2 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Sudden death NOS (General disorders) | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Immune system disorders-Other (Immune system disorders) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 2 | 1
Joint infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 5 | 5
Sepsis (Infections and infestations) | 2 | 7 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Cardiac troponin I increased (Investigations) | 1 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Fibrinogen decreased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3 | 3
Platelet count decreased (Investigations) | 1 | 5 | 2
White blood cell decreased (Investigations) | 0 | 4 | 3
Acidosis (Metabolism and nutrition disorders) | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 4 | 2
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=25) | Azacitidine + Nivolumab (N=25) | Azacitidine +Midostaurin (N=23)
Anemia (Blood and lymphatic system disorders) | 13 | 12 | 13
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 1 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3 | 6
Cardiac disorders-Other (Cardiac disorders) | 1 | 1 | 3
Heart failure (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Blurred vision (Eye disorders) | 0 | 1 | 2
Eye disorders-Other (Eye disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 6
Constipation (Gastrointestinal disorders) | 13 | 7 | 17
Diarrhea (Gastrointestinal disorders) | 6 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 4
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 4 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 3 | 3
Nausea (Gastrointestinal disorders) | 9 | 6 | 12
Oral pain (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2 | 11
Chills (General disorders) | 2 | 1 | 4
Edema limbs (General disorders) | 4 | 4 | 5
Fatigue (General disorders) | 12 | 8 | 15
Fever (General disorders) | 5 | 2 | 2
Gait disturbance (General disorders) | 0 | 2 | 1
General disorders and administration site conditio (General disorders) | 0 | 1 | 2
Injection site reaction (General disorders) | 1 | 4 | 2
Malaise (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 4
Pain (General disorders) | 3 | 2 | 8
Infections and infestations-Other (Infections and infestations) | 3 | 3 | 3
Lung infection (Infections and infestations) | 2 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 2
Skin infection (Infections and infestations) | 2 | 2 | 2
Upper respiratory infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 3
Bruising (Injury, poisoning and procedural complications) | 6 | 2 | 7
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 4
Injury, poisoning and procedural complications-Oth (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 8 | 5 | 7
Alkaline phosphatase increased (Investigations) | 6 | 4 | 9
Aspartate aminotransferase increased (Investigations) | 8 | 7 | 7
Blood bilirubin increased (Investigations) | 4 | 4 | 8
Cardiac troponin I increased (Investigations) | 2 | 1 | 2
Creatinine increased (Investigations) | 6 | 10 | 10
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 4
INR increased (Investigations) | 0 | 2 | 2
Lymphocyte count decreased (Investigations) | 9 | 11 | 9
Neutrophil count decreased (Investigations) | 12 | 10 | 13
Platelet count decreased (Investigations) | 12 | 11 | 13
Serum amylase increased (Investigations) | 0 | 3 | 0
Weight loss (Investigations) | 2 | 4 | 7
White blood cell decreased (Investigations) | 18 | 13 | 15
Anorexia (Metabolism and nutrition disorders) | 4 | 12 | 10
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 9 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 5 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 11 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 4 | 7 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 14 | 9 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 8
Neoplasms benign, malignant and unspecified (incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 3 | 4 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 4
Headache (Nervous system disorders) | 2 | 2 | 6
Lethargy (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 5
Confusion (Psychiatric disorders) | 0 | 3 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 3 | 0 | 5
Insomnia (Psychiatric disorders) | 2 | 3 | 5
Hematuria (Renal and urinary disorders) | 2 | 1 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 3
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 6 | 3
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 2 | 2 | 6
Hot flashes (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 4 | 4
Hypotension (Vascular disorders) | 2 | 3 | 7
Thromboembolic event (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03092674/Prot_SAP_000.pdf